CLINICAL TRIAL: NCT02021474
Title: Phase II Study to Assess the Efficacy and Safety of Subcutaneous AGX-201 for Migraine Prophylaxis
Brief Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of Subcutaneous AGX-201 for Migraine Prophylaxis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AgoneX Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGX-201
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Migraine Prophylaxis
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AGX-201 (Experimental): Placebo-controlled Trial to Assess the Efficacy and Safety of Subcutaneous AGX-201 for Migraine Prophylaxis.
  Interventions: Drug: AGX-201
- Evan's solution = phenol 0.4%, isotonic sodium chloride (Placebo Comparator): Placebo-controlled Trial to Assess the Efficacy and Safety of Subcutaneous AGX-201 for Migraine Prophylaxis.
  Interventions: Drug: Subcutaneous placebo (Evan's solution = phenol 0.4%, isotonic sodium chloride).

INTERVENTIONS:
Drug: AGX-201 — Subcutaneous injection
  Arms: AGX-201
Drug: Subcutaneous placebo (Evan's solution = phenol 0.4%, isotonic sodium chloride). — Subcutaneous injection
  Other Names: Placebo
  Arms: Evan's solution = phenol 0.4%, isotonic sodium chloride

SUMMARY:
This is a prospective multi-center, randomized, double-blind, two treatment period, placebo-controlled study in subjects with migraine headache requiring prophylactic treatment. The patients will be randomized to receive either AGH-201 sc or placebo (matching vehicle only) sc for 16 weeks. The safety and efficacy outcome measures will be assessed at selected dosing segments during the 16 week treatment phase and 4 weeks (week 20), 8 weeks (week 24) after the last Injection.

DETAILED DESCRIPTION:
BACKGROUND Migraine headaches affect more than 28 million persons in the United States (Foundation). Approximately 25% of women and 9% of men experience migraine headaches (Rasmussen BK, 1991) (Lipton RB, 1993) (Ramadan NM, 2002). Individuals with migraine headaches lose an average of 4 to 6 working days each year resulting in a total annual loss nationwide of 64 to 150 million workdays. It is estimated that the direct and indirect cost of migraines is nearly $17 billion (Hu XH, 1999) (RK., 1999). Headache is responsible for approximately 2% of all visits to emergency departments (Goldstein JN, 2006).

Migraine headaches are typically described as recurring, unilateral headache with untreated attacks lasting from 4 to 72 hours. The international headache Society Classification of Headaches list the following diagnostic requirements for migraine headache: at least two of the following features: your lateral location, throbbing character, worsening pain with routine activity, and moderate to severe intensity and at least one of the following features: nausea and/or vomiting and photophobia and phonophobia (Society, 1988).

TREATMENT There is no cure for migraine headaches. The treatments for migraine headaches are typically divided into non-pharmacologic and pharmacologic treatments. The non-pharmacologic treatments are designed to target those actions and behaviors known to trigger migraine headaches. The non-pharmacologic treatments include: regular sleep patterns, regular exercise, and the avoidance of known triggers. Triggers for migraine headaches can include: red wine, aged cheeses, exposure to chemical odors i.e. perfumes and cleaners. Non- pharmacologic therapies also include relaxation training, biofeedback, cognitive - behavioral therapy, hypnosis, transcutaneous electrical nerve stimulation, cervical manipulation, and hyperbaric oxygen.

The pharmacologic treatments for migraine headaches are typically divided into abortive therapies and prophylactic therapies. The abortive therapies are usually divided into nonspecific medications used to treat migraines: analgesics/NSAIDS (acetaminophen, aspirin, ibuprofen, naproxen sodium, ketorolac), and narcotic analgesics (meperidine and butorphanol), adjunctive therapy (metoclopramide, prochlorperazine). Migraine specific abortive therapies include ergotamine derivatives (ergotamine, caffeine plus ergotamine, dihydroergotamine) and the Triptans (Sumatriptan, Naratriptan, Rizatriptan, and Zolmitriptan) (Aukerman, 2002). Unlike the abortive therapies, which are taken to treat an existing headache, prophylactic therapies are taken (usually daily) to reduce the frequency and intensity of migraine headaches. Prophylatic, or preventive medications are generally divided into the first-line agents and second-line agents. First-line therapies for migraine prophylaxis in adults include propranolol (Inderal), timolol (Blocadren), amitriptyline, divalproex (Depakote), sodium valproate, and topiramate (Topamax) (Modi & Lowder, 2006). Agents that could be used as second-line therapy for migraine prophylaxis in adults (listed by evidence of effectiveness) include gabapentin (Neurontin), naproxen (Naprosyn) or naproxen sodium (Anaprox), timed-release dihydroergotamine mesylate (DHE-45), candesartan (Atacand), lisinopril (Zestril), atenolol (Tenormin), metoprolol (Toprol XL), nadolol (Corgard), fluoxetine (Prozac), verapamil (Calan), magnesium, vitamin B2 (riboflavin), coenzyme Q10, hormone therapy (estradiol topical gel [Estrogel]), and botulinum toxin type A (Botox) injections (Modi & Lowder, 2006).

PATHOGENESIS OF MIGRAINE Despite extensive research in the area of migraine headaches, the precise pathogenesis of migraine remains unknown. The list of potential candidates for the pathogenesis of migraines is extensive. For many years the excepted pathogenesis of migraine headaches was that they were due to extracerebral vasodilation. This theory proposes that the auras associated with migraine headache were due to an initial vasoconstriction which is followed by a vasodilatation of extracerebral vessels which resulted in the pain of a migraine headache. Others (Blau, 1984) have proposed that migraine is a primary neurological disturbance with secondary vasomotor changes. Migraine is likely a multi-genic condition with a complex pathophysiology in which both central and peripheral components of trigeminal pain pathway play a role in the signs and symptoms. In the past two decades the trigeminal vascular system (TVS) has been proposed as a possible component of migraine attacks. Nitric oxide has also been proposed as a potential mechanism for migraines, supported by the production of typical migraine headaches in migraneurs treated with nitroglycerin (NTG). 5-hydroooxytryptamine (5-HT) has been implicated in migraine pathophysiology. The role for 5-HT metabolism in migraine is supported by a low central 5-HT disposition associated with increase in 5-HT release during an attack (Panconesi, 2008). Weir and Cader (2011) have proposed that channelopaties may play a role in migraine headaches, especially those with a genetic association. Cortical spreading depression has been implicated as a cause for migraine aura (Weir 2011). The Neurogenic inflammation (NI) theory proposes that, vasodilation and plasma protein extravasation in tissue receiving trigeminal innervation occurs when vasoactive peptides are released from nerve endings (Buzzi, 2005). Burstein, et al., 2011 has proposed that peripheral sensitization is a major contributor to hypersensitivity in many painful syndromes including migraine headaches. In this state primary afferent nociceptive neurons exhibit increased responsiveness to external stimuli at the original site of inflammation or injury. A large number of chemical mediators produced at a site of inflammation or tissue injury can promote excitation and sensitization of nociceptors. These chemical mediators include bradykinin, histamine, serotonin (5-HT), and prostaglandins. Cytokines (interleukins 1, 6 and 8 [IL-1, IL-6, IL-8] and tumor necrosis factor alpha [TNF-alpha]) are inflammatory mediators known to promote peripheral sensitization (Burstein, et al., 2011). Central sensitization which occurs in two distinct phases, the initiation phase and the maintenance phase may play a role in migraine headache. This sensitization is mediated by the excitatory amino acid glutamate and neuropeptides such as substance P and neurotrophic factors. The enhanced neuronal excitability in central sensitization involves the phosphorylation of intracellular and extracellular kinases and the enhanced production of cyclooxygenase. The list of chemical mediators involved in the pathogenesis of migraine is extensive. The scientific investigations required to elucidate the exact mechanisms responsible for migraine headaches continues as an important part of ongoing clinical trials.

GLUCOSE METABOLISM AND MIGRAINE The relationship between migraine headaches and hunger is an accepted and well documented phenomenon. Missing meals can precipitate or trigger a migraine in susceptible individuals. Shaw et al., 1977 showed that migraine patients had impaired tolerance to glucose during migraine attacks compared with control studies. There was an elevation of plasma free fatty acid (FFA) levels during the migraine attacks. Growth hormone and cortisol were elevated and insulin was depressed during attacks. Patients with migraine have impaired insulin sensitivity (Rainero, et al., 2005). During the oral glucose tolerance test (OGTT), glucose plasma concentrations were significantly higher in migraineurs than in controls. Insulin sensitivity (measured by ISI-stumvoll and OGIS-180 indexes) was significantly altered in migraine. Cavestro et al. (2007) reported that headache patients had elevated blood glucose levels when compared to controls. They also documented that insulin levels were elevated in migraineurs when compared to control patients and other headache patients. Additional studies are needed to explore the role of impaired glucose metabolism in migraine including the role that glucose metabolism may play in the development of new therapies for migraine.

ROLE OF HISTAMINE IN MIGRAINE In 2003, Gazerani, et al. demonstrated a correlation between migraine, histamine, and immunoglobulin E. Serum samples were collected (for histamine levels and Immunoglobulin E levels) from 70 patients (18 - 58 years) with migraine during an attack and during remission and from 45 healthy volunteers. The migraine patients were divided into two groups according to their history of allergies (60% having a history of allergies and 40% without a history of allergies). Plasma histamine levels were significantly elevated (P ≤ 0.0001) in patients with migraine both during symptom-free periods (Error! Reference source not found.) and during migraine events (Error! Reference source not found.) when compared to the control group.

* RATIONALE FOR THE USE OF STUDY DRUG IN THE TREATMENT OF STUDY DISEASE In 1991, Guerrero, et al. carried out an initial study that provided evidence for the beneficial effects of histamine in migraine prophylaxis (Millan-Guerrero RO, 1999). Their data showed that subcutaneous administration of low doses (1-10 ng) of histamine induced significant relief from migraine symptoms, with no secondary effects. The possible mechanisms of histamine migraine prophylaxis, can be explained by histamine control of mast cells; the antidromic stimulation of trigeminal nerve endings induces the release of substance P and other neuromodulatory peptides, which in turn stimulate the release of histamine from mast cells. In meningeal blood vessels, activation of H1-receptors by histamine, results in vasodilatation and plasma protein extravasation, causing neurogenic inflammation (Akerman S, 2002). Krabbe and Olesen (Krabbe AA, 1980) and Lassen et al. (Lassen LH, 1995) showed that on migrainous subjects, intravenous administration of relatively high doses of histamine (0.5 mg/kg per minute for 20 min) caused an immediate headache during the infusion, followed by a delayed migraine attack which was abolished by pre-treatment with the H1-R antagonist, mepyramine. However, degranulation of mast cells and neuropeptide release from C fiber endings are inhibited by the histamine at low-concentration interaction with H3-receptors (H3-R), and probably reflects a local feedback circuit between C-fiber nerve endings and mast cells, which control neurogenic inflammation (Dimitriadou V, 1994) (Arrang J-M, 1983) (Arrang J-M G. M.-C., 1987) (Placeholder21). Guerrero, et al. proposed that the administration of low doses of histamine, to achieve and maintain low-circulating concentrations, may lead to a selective interaction of histamine with H3-R. Histamine could constitute a new therapeutic drug in migraine prophylaxis that acts by limiting the excessive inflammatory response involved in migraine pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any race, 18 to 65 years of age inclusive.
2. Patients with a history of migraine (with or without aura) according to the Headache Classification Committee of the IHS. Migraine attacks have to have had an onset before age 50 and have to have been present for at least 12 months.
3. Patients with 4-20 qualified migraine attacks per month over the past three months prior to Screening, as well as during the four weeks of the Baseline Phase will be eligible for entry into this study. The interval between two qualified migraine attacks should be at least 24 hours to be counted as distinct migraine attacks. A qualified migraine attack without aura is defined as a headache that lasts 4-72 hours (if untreated or unsuccessfully treated) or if successfully treated. This attack has at least two of the following characteristics: unilateral location, pulsating quality, moderate or severe intensity that inhibits or prohibits daily activities or aggravation by routine physical activities such as walking up stairs. In addition, at least one of the following symptoms must be present during the headache: nausea, vomiting, or photophobia and phonophobia. A qualified migraine attack with aura must fulfill the same criteria as the headache attack, plus have an associated aura as defined by the Migraine Criteria of the Headache Classification Committee of the International Headache Society. An aura alone that requires acute migraine treatment will also be considered a migraine attack.
4. Male and female patients will be eligible for enrollment. Females should be either of non-childbearing potential by reason of surgery, radiation, menopause (one year post onset), or of childbearing potential and practicing a medically acceptable method of contraception (eg, abstinence, a barrier method plus spermicide, or IUD) for at least one month before study randomization and for two months after the end of the study, and have a negative serum B-hCG at Screening. Pregnant and/or lactating females are excluded. Those women using hormonal contraceptives must also be using an additional approved method of contraception (eg, a barrier method plus spermicide, or IUD) starting with the Baseline Phase and continuing throughout the entire study period.
5. Patients who are willing to participate and have provided written informed consent prior to being exposed to any study-related procedures.

Exclusion Criteria:

1. Patients with chronic daily headaches as defined by more than 20 headache days per month on average during the three months prior to Screening,
2. Patients with cluster headaches and other trigeminal autonomic cephalalgias, and other primary headaches (except tension-type headache) and secondary headaches (defined according to the Headache Classification Committee of the IHS 2004),
3. Patients with a history of being non-responsive to more than two classes of adequately conducted, prophylactic migraine treatments (e.g., beta blockers, calcium channel blockers, tricyclics, MAOIs, valproate (divalproex), topiramate, gabapentin),
4. Patients who use the following medications as described:

   * Use of marketed triptans for 12 days or greater per month on average,
   * Use of ergot-containing medications for 12 days or greater per month on average,
   * Use of NSAIDs, acetaminophen, or isometheptene-containing agents for 15 days or greater per month on average,
   * Use of opioids for 12 days or greater per month on average, ￼ - Use of any two or more of the above medications for 15 days or greater per month on average,
5. Patients with clinically significant neurological illness, other than migraine, that, in the opinion of the Investigators, may have the potential of altering pain perception or reporting,
6. Patients with a history of or currently having major psychiatric disorders including schizophrenia, major depressive disorder, or bipolar disorder,
7. Patients with elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) >= 1.5 times the upper limit of normal (ULN),
8. Patients with evidence of significant active hematological disease; White blood cell (WBC) count cannot be <= 2500/μL or an absolute neutrophil count <= 1000/μL.
9. Patients with clinically significant ECG abnormality, including prolonged QTc (Fridericia correction) defined as >= 450 msec for males and >= 470 msec for females,
10. Patients with clinically significant active hepatic disease, cardiovascular, metabolic, respiratory, renal, endocrinological, gastrointestinal diseases, and bacterial or viral infections within 30 days prior to Screening or during the Baseline Phase,
11. Pregnant or lactating females
12. History of transmeridian travel (across >3 time zones) or shift work (defined as permanent night shift or rotating day/night shift work) within the past 2 weeks or anticipates needing to travel (across >3 time zones) at any time during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in monthly migraine days [time frame: baseline and average over Weeks 3-22]. | 4 week intervals over weeks 3-22
  Mean change from baseline in monthly migraine days [time frame: baseline and average over Weeks 3-22].

SECONDARY OUTCOMES:
Mean change from baseline in monthly migraine days by 4 week intervals [Weeks 3-6, 7-10, 11-14, 15-18, 19-22]. | 4 week time interval
  Mean change from baseline in monthly migraine days by 4 week intervals [Weeks 3-6, 7-10, 11-14, 15-18, 19-22].
Mean Change from Baseline in Monthly Migraine Index (MMI) | Baseline and average over observation period (weeks 3-22)
  Mean Change from Baseline in Monthly Migraine Index (MMI) [ Time Frame: baseline and average over observation period (Weeks 3-22).
  Monthly Migraine Index (MMI):
  Migraine headaches are assigned a number based on the peak intensity of that migraine headache:
  * 1 for a mild migraine headache
  * 2 for a moderate migraine headache
  * 3 for a severe migraine headache.
  The MMI is calculated as follows:
  MMI= Sum of [(Migraine Peak Intensity Level (1-3)) x (Migraine Duration (hours))] / (Distinct Number of Migraine Headaches for that 4 week period)
  Sample Calculation:
  The patient experiences 3 migraine headaches (M1, M2, and M3) in 4 weeks . M1: Intensity Level 3, Duration is 7 hrs M2: Intensity Level 2, Duration 3 hrs M3: Intensity Level 3, Duration 15 hrs MMI= (3x7 + 2x3 + 3x15) / 3 = 24
Mean change from baseline in monthly number of migraines | Baseline and over weeks 3-22
  Mean change from baseline in monthly number of migraines [time frame: baseline and over Weeks 3-22].
Mean change from baseline in monthly number of migraines | 4 week intervals [Weeks 3-6, 7-10, 11-14, 15-18, 19-22].
  Mean change from baseline in monthly number of migraines by 4 week intervals [Weeks 3-6, 7-10, 11-14, 15-18, 19-22].

REFERENCES:
- [Result] Millan-Guerrero RO, Isais-Millan R. [New therapeutic alternatives in migraine prophylaxis using histamine H3 receptor agonists]. Gac Med Mex. 2008 Jul-Aug;144(4):291-5. Spanish. PMID 18942262
- [Result] Millan-Guerrero RO, Isais-Millan S, Barreto-Vizcaino S, Rivera-Castano L, Rios-Madariaga C. Subcutaneous histamine versus botulinum toxin type A in migraine prophylaxis: a randomized, double-blind study. Eur J Neurol. 2009 Jan;16(1):88-94. doi: 10.1111/j.1468-1331.2008.02352.x. PMID 19087155
- [Result] Millan-Guerrero RO, Isais-Millan R, Barreto-Vizcaino S, Gutierrez I, Rivera-Castano L, Trujillo-Hernandez B, Baltazar LM. Subcutaneous histamine versus topiramate in migraine prophylaxis: a double-blind study. Eur Neurol. 2008;59(5):237-42. doi: 10.1159/000115637. Epub 2008 Feb 8. PMID 18264012
- [Result] Millan-Guerrero RO, Isais-Millan R, Barreto-Vizcaino S, Rivera-Castano L, Garcia-Solorzano A, Lopez-Blanca C, Membrila-Maldonado M, Munoz-Solis R. Subcutaneous histamine versus sodium valproate in migraine prophylaxis: a randomized, controlled, double-blind study. Eur J Neurol. 2007 Oct;14(10):1079-84. doi: 10.1111/j.1468-1331.2007.01744.x. PMID 17880560
- [Result] Millan-Guerrero RO, Isais-Millan R, Benjamin TH, Tene CE. Nalpha-methyl histamine safety and efficacy in migraine prophylaxis: phase III study. Can J Neurol Sci. 2006 May;33(2):195-9. doi: 10.1017/s0317167100004960. PMID 16736729
- [Result] Millan Guerrero R, Trujillo Hernandez B, Tene CE. [Subcutaneous histamine in migraine prophylaxis. Initial effects and long-term outcome]. Neurologia. 2006 Mar;21(2):55-9. Spanish. PMID 16525910